CLINICAL TRIAL: NCT05228587
Title: Indocyanine Green Clearance Test in Liver Transplantation: Defining Cut-off Levels for Graft Viability Assessment During Organ Retrieval and for the Prediction of Post-transplant Graft Function Recovery
Brief Title: Indocyanine Green Clearance Test in Liver Transplantation (LivInG)
Acronym: LivInG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Azienda Policlinico Umberto I (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3656
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-01

CONDITIONS: Hepatic and Hepatobiliary Disorders
Keywords: Organ donation; Indocyanine Green Clearance; Liver injury, repair; Liver ischemia-reperfusion injury; Liver dysplasia and pre-neoplasia; Liver Transplant
MeSH Terms: conditions — Digestive System Diseases | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Liver Transplants (Experimental): Indocyanine Green will be injected in liver donors for measuring plasma disappearance rate with a non invasive measurement device.
  Liver recipients will receive indocyanine green injection for measuring plasma disappearance rate at different time-points.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Indocyanine green will be injected in all donor
  Other Names: Injection of Indocyanine green

SUMMARY:
The gap between patients awaiting and those undergoing liver transplantation (LT) continues to grow. Marginal organs carry higher risk of failure after LT however they are increasingly used to fill such gap. Viability assessment of the graft is essential to lower the risk of LT failure and need for emergency re-LT, however this still relies mainly on surgeon's experience. Post-LT graft function recovery assessment is also essential to aid physicians in the management of LT recipients and guide them through challenging decision-making.

With the present study we aim to validate the use of indocyanine green clearance test (IGT) in two settings: in the donor as an objective tool to assess graft viability; in the recipient to assess graft function recovery after LT.

The implementation of IGT in routine practice translates into two main advantages: to avoid using grafts with no chance of recovery and to optimize resource allocation to LT recipients depending on their graft function recovery.

DETAILED DESCRIPTION:
Liver transplantation (LT) is the gold standard treatment for end-stage liver diseases. The success of LT and the expansion of medical conditions that are successfully treated with LT, has caused a growing gap between available organs and patients still dying while awaiting a transplantable organ. Various attempts at fulfilling the gap continue to be made, including donation from live donors, split livers, and utilization of "marginal" deceased donors (e.g. elderly donors, steatotic grafts, donors after cardiac death, etc.). Marginal grafts carry an increased risk of post-transplant failure which is difficult to quantify. Yet, we rely on the donor surgeon's evaluation based on experience. In selected cases, a liver biopsy can be used, however the limitations of liver biopsies in graft viability assessment are well known and extensively questioned in the scientific literature, to the point of being used only in few selected cases by many transplant units. The adoption of an objective measure of graft viability is highly desirable to prevent from transplanting organs at high risk of failure. Similarly, the recovery of organ function after LT is not measured by means of an objective test. This is mainly monitored with laboratory tests, in some cases measuring bile production, and monitoring the clinical evolution of patients condition.

Indocyanine green clearance test (IGT) has been evaluated as a prognostic marker in patients with advanced cirrhosis or awaiting liver transplantation. In addition, it is used as a marker of portal hypertension in cirrhotic patients, as a prognostic factor in intensive care units and is commonly used as part of the preoperative work-up before liver resections. Indocyanine green is administered intravenously, up-taken almost exclusively by hepatocytes and excreted unprocessed in the bile ducts. The disappearance rate from the bloodstream is measured either on a blood sample (i.e. retention rate 15 minutes after injection) or - more recently - with a pulsidensitometric method (i.e. plasma disappearance rate). Slower plasma disappearance rate (PDR) correlate with worse liver function. A cut-off PDR level of >14%/min has been reported to allow safe major liver resections.

The role of IGT in LT has not been investigated extensively yet, in particular for the assessment of graft viability during donation. A correlation between graft steatosis and IGT in the donor has been observed whilst an increased incidence of graft failure has been reported with PDR<11%/min. Conversely, there is more evidence in the recipient setting, with IGT correlating with the occurrence of post-LT complications (PDR cut-off level for increased risk of post-LT complications of <12.85%/min or graft loss and/or patient death of <9.6%/min). However, a correlation between the changes in the values (i.e. the slope) of IGT and graft function recovery has not been studied yet. Since recent technology enables PDR to be measured non-invasively at the bedside, this parameter is an attractive addition to liver function assessment. However, the current state-of-the-art as concerns this technology remains at a low level of evidence and thorough assessment is required.

Hyphotesis and Significance:

We hypothesize to identify an IGT cut-off level to aid the retrieval surgeon in the decision-making process of accepting an organ to be used for LT. Secondly, we hypothesize to identify a correlation between IGT values and post-transplant organ function recovery.

Specific Aim 1:

To identify IGT PDR cut-off level below which the liver graft is not to be used for solid organ transplantation.

Specific Aim 2:

To identify IGT cut-off level(s) below which post-LT organ recovery is impaired (early allograft dysfunction). IGT will be measured at different time-points post-LT: during the anhepatic phase, post-reperfusion, on day 1, 3 and 7. Each time-point measurement will be analyzed for correlation with early allograft dysfunction (EAD). To define distinct classes of risk of early allograft dysfunction based on the slope of IGT values, starting from the donor IGT, ending on day 7 post-LT.

Experimental Design Aim 1:

Organ donors will be managed according to the Italian National Transplant Center (CNT) policy and the current study will not require any change to standard practice. Indocyanine green 20 ml will be administered to the multiorgan donor upon arrival in the operating room by a researcher of this study. The IGT plasma disappearance rate will be measured using the pulsidensitometric method (LiMON System, Impulse Medical System, Munich, Germany - or alternative/equivalent device) by the same researcher, recorded and secured inside a specially designed "IGT Study Box". The value obtained will not be revealed to the surgical retrieval team who will carry out the operation without any deviation from standard practice because of the current study (i.e. surgical team blinded).

Considering our current discard rate of 30% of liver grafts at the time of organ retrieval during 2017 and 2018 years, we expect a discard rate of 40% for organs with an IGT value inferior to 13%/min (cut-off value was chosen from existing literature) and a discard rate of 20% for organs with a IGT value equal to or above 13%/min.

Power calculation for Aim 1:

162 organ retrieval procedures are required for achieving 80% power (alfa 0.05).

Our current activity ranges between 60 and 70 organ retrievals per year and we plan to complete the enrollment in 30-32 months.

Interim analysis once 50% enrollment is complete will be carried out to compare hypothesis (IGT cut-off level <13%/min for liver graft viability) with actual results. Study sample size might be amended accordingly.

Liver transplantation will take place as per our standard protocol and IGT PDR will be measured with the pulsidensitometric method at different time-points:

* T.0(zero): during the anhepatic phase (at completion of total hepatectomy) to calculate potential disappearance of indocyanine green via non-hepatic mechanisms (mainly extravasation in the interstitium as known from available literature). The anhepatic disappearance rate will serve as a correction factor of IGT values until the recipient has evidence of fluid overload >10 L from their pre-LT weight;
* T.LT: after hemodynamic stability is obtained for at least one hour (usually after completion of bile duct reconstruction).
* Measurement of IGT will take place also after 24 hours (T.1) from LT and then on day 3 (T.3) and day 7 (T.7) after LT.

All post-LT IGT values will be recorded on the patient's chart and will be accessible to the clinical staff managing the patient.

LT recipients will receive special informed consent to participate in the study and a dedicated leaflet will be produced to inform patients regarding study aims, possibility to withdraw from the study at any time, possible side effects related to indocyanine green and no financial implication neither for the patient nor for the researchers.

Statistical analyses: for the descriptive analyses, continuous variables will be presented as the medians plus interquartile ranges, and categorical variables will be presented as percentages and frequencies. The Kolmogorov-Smirnov test will be used to verify a normal distribution.

For Aim 1: The study groups (divided depending on IGT values) will be compared using the Mann-Whitney U test for continuous variables; Fisher's exact test will be used for categorical variables. To identify the independent risk factors associated with donor acceptance, a univariate logistic regression analysis will be conducted. Variables with a P value of <0.20 in the univariate analysis will be included in the multivariate logistic regression analysis via the forward stepwise method; the results will be presented as odds ratios (ORs) with 95% confidence intervals (CIs). Receiver operating characteristic (ROC) curves will be plotted for identifying the best IGT threshold value for the diagnosis of donor refusal. Cut-off values will be measured using the highest Youden index (specificity + sensitivity - 1) obtained from the ROC curves.

For Aim 2: descriptive statistics as per Aim 1. In addition, to identify the independent risk factors associated with early allograft dysfunction (EAD), a univariate logistic regression analysis will be conducted. Variables with a P value of <0.20 in the univariate analysis will be included in the multivariate logistic regression analysis via the forward stepwise method; the results will be presented as odds ratios (ORs) with 95% confidence intervals (CIs). Receiver operating characteristic (ROC) curves will be plotted for identifying the best IGT threshold value for the diagnosis of EAD.

Cut-off values will be measured using the highest Youden index (specificity + sensitivity - 1) obtained from the ROC curves.

All patients will be followed until death, graft failure, or last known follow-up visit. Graft survival will be analyzed using the Kaplan-Meier method, and group comparisons will be conducted using the log-rank test. Statistical analyses will be performed using the Statistical Package for the Social Science (SPSS) 22.0 (IBM, USA). All P values will be two-tailed, and P<0.05 will be considered to indicate significance.

Expected outcomes:

* We expect to validate the use of IGT in the setting of organ retrieval to aid the retrieval surgeon in the decision-making process of accepting a liver graft for solid organ transplantation. This will expand the yet limited armamentarium of the retrieval surgeon for graft viability assessment.
* We expect to identify cut-off levels of IGT at distinct time points after LT which could predict the development of EAD or graft failure. In addition, we expect to describe risk classes for the development of EAD by evaluating the slope of IGT from the time of organ retrieval to day 7 post-LT. With this, we will add an objective measure of liver function post-LT to better detect EAD not only by laboratory data or clinical observation, thus offering a useful tool to the transplant physicians managing complex clinical scenarios where there is uncertainty regarding lack of graft function recovery. Undiagnosed EAD or graft failure can lead to delayed indication for re-LT and recipient's death due to overcoming complications.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive liver donors included in the study period
* All consecutive liver recipients transplanted in the study period from a donor tested with Indocyanine Green

Exclusion Criteria:

* Donor or recipients history of allergy to hyodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
To identify IGT PDR cut-off level below which the liver graft is not to be used for solid organ transplantation | During organ donor retrieval surgery
  Organ donors will be managed according to the Italian National Transplant Center (CNT) policy and the current study will not require any change to standard practice. Indocyanine green 20 ml will be administered to the multiorgan donor upon arrival in the operating room by a researcher of this study. The IGT plasma disappearance rate will be measured using the pulsidensitometric method (LiMON System, Impulse Medical System, Munich, Germany - or alternative/equivalent device) by the same researcher, recorded and secured inside a specially designed "IGT Study Box". The value obtained will not be revealed to the surgical retrieval team who will carry out the operation without any deviation from standard practice because of the current study (i.e. surgical team blinded).

SECONDARY OUTCOMES:
To identify IGT PDR cut-off level(s) below which post-LT organ recovery is impaired (early allograft dysfunction). | From Transplant to the 7th postoperative day
  IGT will be measured at different time-points post-LT: during the anhepatic phase, post-reperfusion, on day 1, 3 and 7. Each time-point measurement will be analyzed for correlation with early allograft dysfunction (EAD).
  To define distinct classes of risk of early allograft dysfunction based on the slope of IGT values, starting from the donor IGT, ending on day 7 post-LT.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo IJ, Lefkowitch JH, Feirt N, Alkofer B, Kin C, Samstein B, Guarrera JV, Renz JF. Utility of liver allograft biopsy obtained at procurement. Liver Transpl. 2008 May;14(5):639-46. doi: 10.1002/lt.21419. PMID 18324657
- [Background] Levesque E, Martin E, Dudau D, Lim C, Dhonneur G, Azoulay D. Current use and perspective of indocyanine green clearance in liver diseases. Anaesth Crit Care Pain Med. 2016 Feb;35(1):49-57. doi: 10.1016/j.accpm.2015.06.006. Epub 2015 Oct 21. PMID 26477363
- [Background] Lau H, Man K, Fan ST, Yu WC, Lo CM, Wong J. Evaluation of preoperative hepatic function in patients with hepatocellular carcinoma undergoing hepatectomy. Br J Surg. 1997 Sep;84(9):1255-9. PMID 9313707
- [Background] Wang W, Zhao Q, Hu A, He X, Zhu X. Application of Indocyanine Green (ICG) Detection in Evaluating Early Prognosis in Patients with Fatty Liver Disease After Liver Transplantation. Ann Transplant. 2017 Apr 11;22:208-214. doi: 10.12659/aot.901277. PMID 28396579
- [Background] Tang Y, Han M, Chen M, Wang X, Ji F, Zhao Q, Zhang Z, Ju W, Wang D, Guo Z, He X. Donor Indocyanine Green Clearance Test Predicts Graft Quality and Early Graft Prognosis After Liver Transplantation. Dig Dis Sci. 2017 Nov;62(11):3212-3220. doi: 10.1007/s10620-017-4765-x. Epub 2017 Sep 20. PMID 28932926
- [Background] Levesque E, Saliba F, Benhamida S, Ichai P, Azoulay D, Adam R, Castaing D, Samuel D. Plasma disappearance rate of indocyanine green: a tool to evaluate early graft outcome after liver transplantation. Liver Transpl. 2009 Oct;15(10):1358-64. doi: 10.1002/lt.21805. PMID 19790157
- [Background] Schneider L, Spiegel M, Latanowicz S, Weigand MA, Schmidt J, Werner J, Stremmel W, Eisenbach C. Noninvasive indocyanine green plasma disappearance rate predicts early complications, graft failure or death after liver transplantation. Hepatobiliary Pancreat Dis Int. 2011 Aug;10(4):362-8. doi: 10.1016/s1499-3872(11)60061-1. PMID 21813383
- [Background] Imamura H, Sano K, Sugawara Y, Kokudo N, Makuuchi M. Assessment of hepatic reserve for indication of hepatic resection: decision tree incorporating indocyanine green test. J Hepatobiliary Pancreat Surg. 2005;12(1):16-22. doi: 10.1007/s00534-004-0965-9. PMID 15754094
- [Background] Olthoff KM, Kulik L, Samstein B, Kaminski M, Abecassis M, Emond J, Shaked A, Christie JD. Validation of a current definition of early allograft dysfunction in liver transplant recipients and analysis of risk factors. Liver Transpl. 2010 Aug;16(8):943-9. doi: 10.1002/lt.22091. PMID 20677285
- [Derived] Coppola A, Bianco G, Lai Q, Marrone G, Caimano M, Agnes S, Spoletini G. Indocyanine green clearance test in liver transplantation: defining cut-off levels for graft viability assessment during organ retrieval and for the prediction of post-transplant graft function recovery - the Liver Indocyanine Green (LivInG) Trial Study Protocol. BMJ Open. 2022 Aug 1;12(8):e063081. doi: 10.1136/bmjopen-2022-063081. PMID 35914905